CLINICAL TRIAL: NCT04763915
Title: Improving Care After Inherited Cancer Testing (IMPACT) Study
Brief Title: Improving Care After Inherited Cancer Testing
Acronym: IMPACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of South Florida (Other)
Responsible Party: Principal Investigator, Tuya Pal, Associate Director for Cancer Health Disparities, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VICC SUPP 2112; U01CA254832 (NIH)
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Inherited Cancer Syndrome; Prostate Cancer; Colorectal Cancer; Endometrial Cancer; Breast Cancer
Keywords: Inherited Cancer Gene; Pathogenic/Likely Pathogenic Variant; Variant of Uncertain Significance; Cancer Risk Management; Family Sharing
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary; Prostatic Neoplasms; Colorectal Neoplasms; Endometrial Neoplasms; Breast Neoplasms | interventions — Surveys and Questionnaires; Interviews as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GeneSHARE (Experimental): Access to GeneSHARE, a web-based toolkit including interactive and narrative components to enhance FC of genetic test results.
  Interventions: Other: Correlative Studies (Survey); Other: Correlative Studies (Interview); Behavioral: GeneSHARE
- LivingLabReport (Experimental): Access to LivingLabReport, a website containing multiple resources including a summary of the patient's genetic test results, condition-specific information, recommended CRM, and information on accessing CRM services.
  Interventions: Other: Correlative Studies (Survey); Other: Correlative Studies (Interview); Behavioral: LivingLabReport
- Standard-of-care (Active Comparator): Receive standard-of-care from their treating healthcare provider.
  Interventions: Other: Correlative Studies (Survey); Other: Correlative Studies (Interview); Behavioral: Standard-of-care & Adaptive Intervention
- Variants of Uncertain Significance (VUS) Pilot Study (Experimental): Participants are provided access to VUS educational resources including video and written education and assistance for speaking with family members.
  Interventions: Other: Correlative Studies (Survey); Other: Access to Education Materials

INTERVENTIONS:
Other: Correlative Studies (Survey) — Administer surveys
Other: Correlative Studies (Interview) — In-depth interviews among a subset of participants after the 12-month follow-up survey to either: 1) determine additional resources and tailored message that would be helpful; or 2) assess the adaptive intervention
  Arms: GeneSHARE; LivingLabReport; Standard-of-care
Behavioral: GeneSHARE — Access to GeneSHARE, a web-based toolkit which includes interactive and narrative components to enhance FC of genetic test results.
  Arms: GeneSHARE
Behavioral: LivingLabReport — Access to LivingLabReport, a website containing multiple resources including a summary of the patient's genetic test results, condition-specific information, recommended CRM, and information on accessing CRM services.
  Arms: LivingLabReport
Behavioral: Standard-of-care & Adaptive Intervention — Receive standard-of-care from their treating healthcare provider. A subset of individuals will also be asked to test and pilot the adaptive intervention, which will consist of tailored resources to promote CRM and FC, after the 12-month follow-up survey.
  Arms: Standard-of-care
Other: Access to Education Materials — Receive access to VUS educational materials
  Arms: Variants of Uncertain Significance (VUS) Pilot Study

SUMMARY:
The IMPACT Study seeks to refine and evaluate the effectiveness of interventions on improving guideline-adherent cancer risk management (CRM) and family communication (FC) of genetic test results for individuals with a documented pathogenic/likely pathogenic (P/LP) variant, and FC of family cancer history for individuals with a variant of uncertain significance (VUS) in an inherited cancer gene.

DETAILED DESCRIPTION:
Through recruitment of a racially, geographically, and socioeconomically diverse sample of patients, we will achieve the following aims:

1. Evaluate factors associated with access to genetic risk assessment, counseling, and testing services.
2. Conduct a randomized controlled trial to assess the effectiveness of interventions on improving guideline-adherent CRM and FC of genetic test results among individuals with a P/LP variant in an inherited cancer gene.
3. Conduct a pilot study to assess the effectiveness of an intervention on improving FC of family cancer history among individuals with a VUS in an inherited cancer gene.
4. Create and pilot an adaptive intervention to tailor resources to promote CRM and FC.
5. Document and compare multiple implementation outcomes across the different interventions to maximize their effectiveness and improve reach to underserved populations.

ELIGIBILITY:
Randomized Controlled Trial Eligibility: All trial participants will be autonomous adults who are capable of participating in the study

Inclusion Criteria:

* English-speaking men and women aged 18 years or older
* Not adopted (i.e., have information about their biological relatives)
* Have access to internet and a computer, tablet, or smartphone
* Documented pathogenic/likely pathogenic variant in an inherited cancer gene that has CRM guidelines listed in the National Comprehensive Cancer Network (NCCN) Genetic/Familial Panel focused on Breast, Ovarian, and Pancreatic or Colorectal cancers
* Must meet at least one of the following criteria:

  * Intervention A (GeneSHARE) criteria: Have at least one at-risk adult, living relative who either:

    * has not been told about the genetic test result by the participant
    * has not had their own genetic testing
  * Intervention B (LivingLabReport) criteria: Are non-adherent (i.e., either undertreatment or overtreatment) to at least one of the current NCCN CRM guidelines or if currently adherent, require ongoing cancer screening

VUS Pilot Study Eligibility: All VUS pilot study participants will be autonomous adults who are capable of participating in the study. Eligibility criteria include:

* English-speaking men and women aged 18 years or older
* Not adopted (i.e., have information about their biological relatives)
* Have access to internet and a computer, tablet, or smartphone
* Documented VUS in an inherited cancer gene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 720 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in FC of genetic test results (if P/LP variant result) or family history of cancer (if VUS result) | 12 months
  Having at least one additional at-risk adult, living relative with whom the participant has shared their test result, information about testing, or family history of cancer for the first time or has subsequently followed up with a relative
Change in CRM | 12 months
  Ongoing guideline-adherent CRM or a change towards guideline-adherent CRM per National Comprehensive Cancer Network (NCCN) CRM guidelines based on genetic test results as measured by survey data and verified through medical records where possible and/or appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Tuya Pal, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cragun D, Beckstead J, Farmer M, Hooker G, Dean M, Matloff E, Reid S, Tezak A, Weidner A, Whisenant JG, Pal T. IMProving care After inherited Cancer Testing (IMPACT) study: protocol of a randomized trial evaluating the efficacy of two interventions designed to improve cancer risk management and family communication of genetic test results. BMC Cancer. 2021 Oct 13;21(1):1099. doi: 10.1186/s12885-021-08822-4. PMID 34645413

DOCUMENTS (1):
  • Informed Consent Form (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/15/NCT04763915/ICF_001.pdf